CLINICAL TRIAL: NCT04482283
Title: Epidemiological 2-year Prospective Study to Estimate the Prevalence and Evolution of Heart Failure and Identify Potential Predictors for the Development of Symptomatic HF in Patients withT2 Diabetes Mellitus at High CV Risk
Brief Title: HF Prevalence and Evolution of HF in DM II Patients at High Risk
Acronym: HF-LanDMark
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00313
Record Dates: First submitted 2020-07-20; First posted 2020-07-22 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: RELATED REGISTRY SEARCH

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
This is an epidemiological, single-country, multicenter, 2-year prospective cohort study based on both primary and secondary data collection, which will include a representative sample of 300 eligible T2DM patients managed in real-life settings in Greece. A cross-sectional approach will be applied for addressing the primary objective of the study (prevalence of HF) and for determining potential predictors associated with HF stage and the presence of symptomatic HF at enrollment, whereas the prospective cohort phase will capture the 2-year incidence rate of progression to symptomatic HF as well the long-term outcomes of interest. Τhe study will be conducted and reported as per the Good Pharmacoepidemiology Practice and the local rules and regulations. The study will be carried out by approximately 8 cardiology departments that are HF centers of excellence. In addition, aiming at facilitating recruitment, a referral network will be formed comprising endocrinologists, diabetologists, internists and general practitioners treating DM and practicing at the private healthcare sector or at public health facilities.

The overall study duration is expected to be 51 months, including an 27-month recruitment period and a 24-month observation period per patient. Εach patient will be followed for up to 24 months, or until death, withdrawal of consent, or physician's decision for patient withdrawal, whichever occurs earlier. Follow-up visit frequency will be determined by the participating Investigators, however study-related data will be collected at enrollment and at 6-, 12-, 18-, and 24-month data collection timepoints post-enrollment. Data collection at enrollment, and at 6 and 24 months post-enrollment will be performed in the context of on-site routine clinical visits at the hospital sites whereas data collection at 12 and 18 months will be performed through telephone contacts.

DETAILED DESCRIPTION:
Background/Rationale:

Heart failure (HF) is a major contributor to cardiovascular morbidity and mortality, and one of the most common urgent cardiovascular (CV) presentations in patients with diabetes mellitus (DM). The incidence of HF is higher in adults with DM than in those without. In addition, among patients with HF, those diagnosed with DM have a higher risk of CV death or hospitalization for HF (HHF). As a result of the intersection of DM, atherosclerotic CV disease, and HF, the importance of determining diabetes therapies that are not only safe but also effective in reducing CV risk is paramount. Recently, three large randomized trials have shown that sodium-glucose transport protein 2 (SGLT2) inhibitors, used for the treatment of DM, significantly reduced the risk for HHF. In addition, recent evidence indicates the beneficial effects of the SGLT2 inhibitor dapagliflozin in terms of reducing the risk of worsening HF or CV-related death in patients with established HF and a reduced ejection fraction, regardless of the presence or absence of DM.

As per the American College of Cardiology/American Heart Association (ACC/AHA), patients with DM have at least stage A HF; thus, early identification of patients at higher risk and prompt intervention with medical treatments may not only provide symptomatic relief but also delay the development of HF. In view of the scarce epidemiological data regarding the classification of HF stages among diabetics and the fact that imaging and circulating biomarkers could be of significant prognostic value, there is an eminent need for comprehensive phenotypic characterization of high-risk patients that could provide valuable insight to support the optimal care transition and timely referral of patients with unrecognized HF who fit a particular profile to HF specialists for appropriate diagnostic evaluation and planning of optimal treatment and follow-up care. In light of the above, this epidemiological study aims to generate novel real-world data on the prevalence and evolution of HF stages as well as to explore potential determinants of the development of symptomatic HF, among patients diagnosed with type 2 DM (T2DM) in the past 5 years who are at high CV risk, in Greece. This study, complemented with cardiac imaging and circulating biomarkers data, could provide the necessary data for the creation of an algorithm for the selection of a high-risk population that could draw a greater benefit from medical interventions. Furthermore, the study will attempt to measure the burden of HF- and CV-related healthcare resource utilisation (HCRU) by HF stage and to capture the impact of symptomatic HF on patient-perceived health status.

Objectives and Hypotheses:

The study is not planned to reject or affirm any formal statistical hypothesis. It is noted that the term 'overall study population' used in the objectives below encompasses high CV risk T2DM patients undiagnosed with HF at study enrollment who fulfil the study eligibility criteria.

Primary Objective The primary objective of this study is to estimate the prevalence of previously undiagnosed, symptomatic (clinically overt) HF and to determine the distribution of HF stages (as defined by the ACC/AHA classification) in the overall study population and by New York Heart Association (NYHA) functional classification.

Secondary Objectives

* To assess the evolution of HF stages and of the severity of functional limitation imposed by HF (as assessed by NYHA classification) over the 2-year observation period in the overall study population and by HF stage at enrollment.
* To estimate the incidence of symptomatic HF over the 2-year observation period in the study subpopulation with preclinical HF (Stages A and B) at enrollment.
* To estimate the rate of progression from asymptomatic left ventricular dysfunction (Stage B) at enrollment to symptomatic HF, in the study subpopulation with HF Stage B at enrollment.
* To characterize the baseline clinical, biochemical and echocardiographic profile in the overall study population and by HF stage at enrollment.
* To capture the patient-perceived impact of HF on health status (symptoms, function, and quality of life) and to measure the change in health status from enrollment at 6 and 24 months post-enrollment using the short version of the HF-specific Kansas City Cardiomyopathy Questionnaire (KCCQ-12) in the study subpopulation diagnosed with symptomatic HF (Stage C) at enrollment.
* To assess the HF- and CV-related HCRU in terms of inpatient and outpatient healthcare encounters and use of medical procedures/interventions/tests over the 2-year observation period in the overall study population and by HF stage at enrollment.

Exploratory Objectives

* To identify which baseline clinical, echocardiographic and biochemical parameters of interest are associated with the HF stage at enrollment and to determine potential predictors of symptomatic HF.
* To identify baseline clinical, echocardiographic and biochemical parameters that are associated with progression from preclinical to symptomatic HF, in the study subpopulation with preclinical HF at enrollment.
* To explore whether the change in NT-proBNP level from enrollment to 6 months can serve as a possible predictor for HF- and CV-related morbidity and mortality outcomes in the overall study population.
* To identify number of patients who experience an acute kidney injury event
* To explore changes in eGFR during the study observation period

Methods:

Study design:

This is an epidemiological, single-country, multicenter, 2-year prospective cohort study based on both primary and secondary data collection, which will include a representative sample of 300 eligible T2DM patients managed in real-life settings in Greece. A cross-sectional approach will be applied for addressing the primary objective of the study (prevalence of HF) and for determining potential predictors associated with HF stage and the presence of symptomatic HF at enrollment, whereas the prospective cohort phase will capture the 2-year incidence rate of progression to symptomatic HF as well the long-term outcomes of interest. Τhe study will be conducted and reported as per the Good Pharmacoepidemiology Practice and the local rules and regulations. The study will be carried out by approximately 8 cardiology departments that are HF centers of excellence. In addition, aiming at facilitating recruitment, a referral network will be formed comprising endocrinologists, diabetologists, internists and general practitioners treating DM and practicing at the private healthcare sector or at public health facilities.

The overall study duration is expected to be 51 months, including an 27-month recruitment period and a 24-month observation period per patient. Εach patient will be followed for up to 24 months, or until death, withdrawal of consent, or physician's decision for patient withdrawal, whichever occurs earlier. Follow-up visit frequency will be determined by the participating Investigators, however study-related data will be collected at enrollment and at 6-, 12-, 18-, and 24-month data collection timepoints post-enrollment. Data collection at enrollment, and at 6 and 24 months post-enrollment will be performed in the context of on-site routine clinical visits at the hospital sites whereas data collection at 12 and 18 months will be performed through telephone contacts.

Data Source(s):

Data collection will be carried through a web-based data capture system (eCRF). Primary data -which will be obtained at enrollment and prospectively during the study visits/contacts as performed per standard clinical practice or through patient self-report- will mainly be employed. Data regarding the patient-perceived health status will be collected through completion of the KCCQ-12 instrument at enrollment and at 6 and 24 months post-enrollment. Data regarding the patient's medical, DM- and CV-related history will be abstracted from patients' medicals records and patient self-report, where applicable. Clinical decisions concerning the optimum diabetes, HF and CV risk management strategy for a particular patient are taken independently of and/or prior to any decision by the physician to invite a patient to participate in the study. The medications administered for T2DM, HF, CV diseases and any underlying CV risk factors will be recorded and presented only by drug classes.

ELIGIBILITY:
Inclusion Criteria:

* Female or male outpatients aged 40 to 80 years (inclusive) at the time of providing informed consent.
* T2DM diagnosis within 10 years prior to enrollment.
* Patients must have a high or very high cardiovascular risk (as outlined in 2019 ESC Guidelines on diabetes, pre-diabetes and CV diseases).

Note: Very high CV risk is defined as having either established CV disease, or other target organ damage (proteinuria, LVH, or retinopathy), or at least three major risk factors. High CV risk is defined as age ≥ 50 years and presence of at least one additional major risk factor. Major risk factors include age ≥ 50 years, hypertension, dyslipidemia, smoking, and obesity.

* Patients must have available medical records for data abstraction to meet the objectives of the study.
* Written signed and dated informed consent.

Exclusion Criteria:

* Diagnosis of type 1 DM.
* Treatment with SGLT2 inhibitor at the time of providing informed consent.
* History of HF (defined as current or previous receipt of treatment prescribed for the management of HF, and/or hospitalization for HF at any time in the past).
* Patients with limitations in their functional capacity that, as per the physician's judgment, are attributed to non-cardiac medical reason or condition (such as lung disease, musculoskeletal disorders, infection, endocrine disorders etc.).
* History of any malignancy within the 5-year period prior to enrollment (with the exception of successfully treated non-melanoma skin cancers).
* Chronic cystitis and/or recurrent genital or urinary tract infections (3 or more in the last year).
* Acute kidney injury or rapidly progressing renal disease.
* Severe renal impairment (estimated glomerular filtration rate [eGFR] <30 mL/min/1.73m2 using the CKD-EPI equation).
* Hematuria (confirmed by microscopic evaluation) with no explanation as judged by the study physician.
* HbA1c level ≥12%.
* Aspartate or alanine aminotransferase >3 x upper limit of normal (ULN) or total bilirubin >2.5xULN.
* Pregnant or breastfeeding patient.
* Patients with lifetime expectancy less than 2 years due to any non-cardiovascular cause or with any non-cardiac condition which, in the judgment of the Investigator, may render the patient unable to complete the study.
* Patients who are currently receiving treatment with any investigational drug/device/intervention or have received any investigational product within 1 month or 5 half-lives of the investigational agent (whichever is longer) prior to enrollment.
* Patients who have already been enrolled in this study or in a study of the same design which the physician has good reasons to believe that it is this study (to exclude enrollment of the same patient by two different sites).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the study encompasses high CV risk T2DM patients undiagnosed with HF at study enrollment who fulfil the study eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
Proportion of patients diagnosed with symptomatic HF | 2 years
  Proportion of patients diagnosed with symptomatic HF (Stage C) at enrollment in the overall study population

CONTACTS AND LOCATIONS:
Overall Officials: IOANNIS PARISSIS, Principal Investigator — AZ Greece
Locations (6):
- Greece (6):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Larissa
  - Research Site, Pátrai
  - Research Site, Thessaloniki

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Parissis J, Georgiou C, Bistola V, Karavidas A, Vassilikos VP, Kanakakis J, Davlouros P, Tziakas DN, Alexanian IP, Kochiadakis G, Triposkiadis F, Karvounis H, Gourlis D, Papoutsidakis N, Polyzogopoulou E, Vlachopoulos C. Rationale and Design of Heart Failure Prevalence and Evolution of Heart Failure in Diabetes Mellitus Type II Patients at High Risk (HF-LanDMark Study). J Clin Med. 2023 Sep 30;12(19):6319. doi: 10.3390/jcm12196319. PMID 37834963
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1843R00313&attachmentIdentifier=0991f081-c850-4a7e-b160-6ba666d873c3&fileName=D1843R00313_Redacted_CSR_Synopsis.pdf&versionIdentifier=